CLINICAL TRIAL: NCT05588232
Title: Prospective Randomized Comparative Study Evaluating the Efficacy of Therapeutic Virtual Reality Versus Pharmacological Sedation on Pain and Anxiety During Interventional Cardiology Procedures
Brief Title: the Effectiveness of Therapeutic Virtual Reality Versus Pharmacological Sedation on Pain and Anxiety During Interventional Cardiology Procedures
Acronym: VirtuCardio
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-A01130-41
Record Dates: First submitted 2022-10-18; First posted 2022-10-20 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Virtual Reality; Drug Sedation; Coronarography; Angiography

STUDY DESIGN:
Intervention Model Description: Monocentric, prospective, comparative, randomized, open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient with virtual reality (Experimental): The virtual reality sedation-analgesia solution developed by Deepsen combines 3D environment content with medical hypnosis techniques. The technology includes a wearable visual headset that contains head movement sensors, enabling patient interaction in the virtual environment, as well as isolating headphones.
  Interventions: Procedure: scheduled outpatient interventions in interventional cardiology
- Patient with pharmacological sedation (Active Comparator)
  Interventions: Procedure: scheduled outpatient interventions in interventional cardiology

INTERVENTIONS:
Procedure: scheduled outpatient interventions in interventional cardiology — coronary angiography, coronary angioplasty, peripheral angioplasty (carotid arteries or lower limbs)

SUMMARY:
Immersion sedation in virtual reality could be an alternative to conventional pharmacological sedation, during interventional cardiology acts on pain and anxiety control.

The objective of this study is to determine whether virtual reality immersion is non-inferior to drug sedation on pain and anxiety, during coronary angiography or angioplasty.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* who must benefit from one of the following scheduled interventional cardiology outpatient procedures: coronary angiography, coronary angioplasty, peripheral angioplasty (lower limbs)
* Affiliation to a social security scheme or beneficiary of such a scheme.
* Patient having signed the free and informed consent

Exclusion Criteria:

* Dementia
* Language barrier
* Claustrophobia
* Nausea
* History of intolerance to Virtual Reality
* Patient with epilepsy
* Refusal to participate in the study
* Protected patient: minor, adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision
* Pregnant, breastfeeding or parturient woman
* Unstable patient (state of shock, respiratory or neurological distress)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2021-12-11 (Actual); Study Completion 2022-02-24 (Actual)

PRIMARY OUTCOMES:
Maximum pain during the interventional cardiology procedures | 1 day
  measured on a scale of 0 to 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Claude Bernard, Metz, France